CLINICAL TRIAL: NCT03459469
Title: Phase 1 Trial of BC2059 (Tegavivint) in Patients With Unresectable Desmoid Tumor
Brief Title: Phase I, Open-label, Non-randomized Study to Evaluate Safety of BC2059
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Iterion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCI-001-DT17
Record Dates: First submitted 2018-03-01; First posted 2018-03-09 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Desmoid Tumor
MeSH Terms: conditions — Desmoid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational drug (Experimental): An open-label, non-randomized study to evaluate safety of Tegavivint administered intravenously to subjects with proven primary or recurrent desmoid tumor that is unresectable and symptomatic or progressive.
  Interventions: Drug: Tegavivint

INTERVENTIONS:
Drug: Tegavivint — This is an Investigational drug
  Other Names: BC2059

SUMMARY:
Phase I, open-label, non-randomized study to evaluate safety of BC2059 administered intravenously to subjects with proven primary or recurrent desmoid tumor that is unresectable and symptomatic or progressive.

DETAILED DESCRIPTION:
This study is a phase I, open-label, non-randomized study to evaluate safety of BC2059 administered intravenously to subjects with proven primary or recurrent desmoid tumor that is unresectable and symptomatic or progressive. This study will utilize single patient cohorts for the first two dose levels in order to minimize sub-optimal drug exposures, followed by a conventional 3+3 dose escalation phase to achieve MTD or RP2D determined by pharmacokinetics or biologically relevant activity. Once MTD or RP2D is determined, that dose level cohort will expand to 14 patients enrolled to collect additional safety PK and PD data. If at least 1 patient has clinical benefit, the dose expansion phase will be expanded by a further 11 patients (25 total in at RP2D). The total duration of study for each subject will be dependent upon the safety, tolerability and efficacy of BC2059

ELIGIBILITY:
Inclusion criteria

1. Patients with histologically proven primary or recurrent desmoid tumor with currently bi-dimensionally measurable tumor by WHO criteria.
2. Patients with disease that is either unresectable or for which the patient refuses surgery but is currently progressing, as defined by:

   * 20% increase in tumor volume within 6 months OR
   * Recurrent disease within 1 year of surgery OR
   * Desmoid related symptoms as documented by a PRO questionnaire and documentation that symptoms are related to desmoid and not prior therapies.
3. Willingness to provide tumor biopsies prior to treatment and while on treatment
4. Patients may have been previously treated with local therapies such as surgery, radiation, radiofrequency ablation, or cryosurgery provided this has been completed at least 4 weeks prior to registration and recovered from therapy related toxicity to less than CTCAE grade 2 and show no improvement in tumor size or symptom score.
5. Patients may have been treated with systemic therapies such as tyrosine kinase inhibitors, hormone inhibitors or nonsteroidal anti-inflammatory drugs (NSAIDs) provided this has been completed at least 4 weeks prior to registration and recovered from any therapy related toxicity to less than CTCAE grade 2 and show no improvement in tumor size or symptom score.
6. Patients may have been treated with systemic therapies such as cytotoxics, biologics or other unclassified experimental therapies provided this has been completed at least 8 weeks prior to registration and recovered from any therapy related toxicity to less than CTCAE grade 2 and show no improvement in tumor size or symptom score.
7. Patients who have been treated with immune therapies such as vaccines, dendritic or other whole cell therapies, oncolytic or other viral approaches within the preceding 12 months should be discussed with the Medical Monitor prior to screening and enrollment into the study to determine eligibility.
8. Age: 18 and over (no pre-pubertal patients)
9. ECOG Performance status: 0-1
10. Women of child-bearing potential (WOCBP) and men who are sexually active with WOCBP must agree to use one highly effective method of contraception, including hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy or tubal ligation; and one effective method of contraception, including male condom, female condom, cervical cap, diaphragm or contraceptive sponge or abstain from sex for the duration of study participation and for 4 months following completion of BC2059 administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. See section 8.7.3 for more information.

    Contraception includes:
    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
    * Use of oral (estrogen and progesterone), injected or implanted combined hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    * Sexually active males must use a condom during intercourse while taking drug and for 4 months after stopping study treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

    In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
11. Hematopoietic:

    * Absolute granulocyte count ≥ 1,500/mm3
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin at least 10.0 g/dL (transfusion allowed, subjects that require transfusion or growth factor need to demonstrate stable hemoglobin for at least 7 consecutive days of hemoglobin ≥ 10 g/dL)
12. Hepatic:

    * Bilirubin no greater than 1.5 times institutional upper limit of normal, in the absence of documented Gilbert's syndrome
    * Transaminases no greater than 3 times upper limit of normal (ULN)
    * Alkaline phosphatase no greater than 3 times ULN
13. Renal: Creatinine clearance ≥75 mL/min by Cockcroft-Gault
14. Pulmonary:

    * Diffusing capacity of the lung for carbon monoxide (DLCO) greater than 75% predicted by single breath test
    * Capillary oxygen saturation (O2 sat) > 95% by pulse oximetry

Exclusion Criteria

1. Patients who have not recovered to grade 1 from adverse events related to prior therapy excluding those considered not clinically significant (ex. Lymphopenia).
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to BC2059 or other agents used in study
3. Patients with metabolic bone disease (ex. Hyperparathyroidism, Paget's disease, or osteomalacia)
4. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality or QTc > 480 msec
5. Uncontrolled concurrent illness including, but not limited to: ongoing or active infection (Viral, bacterial, fungal or other)
6. Psychiatric illness/social situations that would limit compliance with study requirements
7. Pregnant and breastfeeding women are excluded from this study. The effects of BC2059 on the developing human fetus have the potential for teratogenic or abortifacient effects. There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BC2059.
8. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with BC2059
9. Patients with abnormal serum chemistry values other than the specific limits detailed above, that in the opinion of the Investigator is considered to be clinically significant, should be discussed with the Medical Monitor before being enrolled in the study.
10. Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples
11. Personal history of malignancy except:

    * Cervical intraepithelial neoplasia;
    * Skin basal cell carcinoma;
    * Treated localized prostate carcinoma with PSA <1 ng/mL;
    * Neoplasia treated with curative intent, in remission for at least five years and considered at low risk of relapse.
12. Patients with familial adenomatous polyposis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability | 12 Months
  Adverse events, Serious adverse events and Dose limiting toxicities

SECONDARY OUTCOMES:
1. To determine the durability of response (DOR) to BC2059 after the achievement of best response | 12 Months
  Assessing CR and PR

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Princess Margaret Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No